CLINICAL TRIAL: NCT03317496
Title: A MULTICENTER, OPEN-LABEL, PHASE 1B/2 STUDY TO EVALUATE SAFETY AND EFFICACY OF AVELUMAB (MSB0010718C) IN COMBINATION WITH CHEMOTHERAPY WITH OR WITHOUT OTHER ANTI-CANCER IMMUNOTHERAPIES AS FIRST-LINE TREATMENT IN PATIENTS WITH ADVANCED MALIGNANCIES
Brief Title: Safety And Efficacy Study Of Avelumab Plus Chemotherapy With Or Without Other Anti-Cancer Immunotherapy Agents In Patients With Advanced Malignancies
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: The study was terminated since there was no need for further safety or efficacy data to be collected. The participants having benefit from the investigational treatments have been moved to a continuation study (NCT05059522).
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: B9991023; B9991023 (Other: Pfizer); 2017-001741-27 (EudraCT Number); JAVELIN CHEMOTHERAPY MEDLEY (Other: Alias Study Number)
Record Dates: First submitted 2017-09-29; First posted 2017-10-23 (Actual); Results first posted 2022-06-23 (Actual); Last update posted 2023-08-29 (Actual); Status verified 2023-08

CONDITIONS: Non-small Cell Lung Cancer; Urothelial Cancer
Keywords: Avelumab, immunotherapy, PD-L1 inhibitor, non-small cell lung cancer (NSCLC), urothelial cancer (UC), carboplatin, pemetrexed, gemcitabine, cisplatin
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — avelumab; Pemetrexed; Carboplatin; Gemcitabine; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Group A Cohort A1 (Experimental): Non-squamous non-small cell lung cancer (NSCLC) patients treated with 800 mg avelumab plus pemetrexed/carboplatin
  Interventions: Drug: Avelumab 800 mg in combination with pemetrexed / carboplatin
- Group A Cohort A2 (Experimental): Cisplatin-eligible urothelial cancer (UC)patients treated with 800 mg avelumab plus gemcitabine/cisplatin
  Interventions: Drug: Avelumab 800 mg in combination with gemcitabine / cisplatin.
- Group A Cohort A3 (Experimental): Non-squamous non-small cell lung cancer (NSCLC) patients treated with 1200 mg avelumab plus pemetrexed/carboplatin
  Interventions: Drug: Avelumab 1200 mg in combination with pemetrexed/carboplatin
- Group A Cohort A4 (Experimental): Cisplatin-eligible urothelial cancer (UC) patients treated with 1200 mg avelumab plus gemcitabine/cisplatin
  Interventions: Drug: Avelumab 1200 mg in combination with gemcitabine/cisplatin

INTERVENTIONS:
Drug: Avelumab 800 mg in combination with pemetrexed / carboplatin — Avelumab Pemetrexed Carboplatin
  Arms: Group A Cohort A1
Drug: Avelumab 800 mg in combination with gemcitabine / cisplatin. — Avelumab Gemcitabine Cisplatin
  Arms: Group A Cohort A2
Drug: Avelumab 1200 mg in combination with pemetrexed/carboplatin — Avelumab Pemetrexed Carboplatin
  Arms: Group A Cohort A3
Drug: Avelumab 1200 mg in combination with gemcitabine/cisplatin — Avelumab Gemcitabine Cisplatin
  Arms: Group A Cohort A4

SUMMARY:
This is a Phase 1b/2, open label, multicenter, safety and clinical activity study of avelumab in combination with chemotherapy as first-line treatment of adult patients with locally advanced or metastatic solid tumors. Initially, avelumab will be evaluated in combination with pemetrexed and carboplatin in patients with advanced non-squamous non-small cell lung cancer (NSCLC) (Cohort A1) and in combination with gemcitabine and cisplatin in patients with cisplatin-eligible urothelial (bladder) cancer (UC) (Cohort A2). As more information is learned about other anti-cancer immunotherapy agents, in future portions of the study, avelumab may be combined with chemotherapy and other anti-cancer immunotherapy agents in patients with these same or different tumor types.

DETAILED DESCRIPTION:
This is a Phase 1b/2, open label, multicenter, safety, clinical activity, pharmacokinetic (PK), and pharmacodynamics (PD) study of avelumab in combination with chemotherapy with or without other anti-cancer immunotherapies, as first-line treatment of adult patients with locally advanced or metastatic solid tumors. Initially, avelumab will be evaluated in combination with pemetrexed and carboplatin in patients with advanced non-squamous non-small cell lung cancer (NSCLC) (Cohort A1) and with gemcitabine and cisplatin in patients with cisplatin-eligible urothelial cancer (UC) (Cohort A2).

Given the growing preclinical and clinical indications that combinations of anti-cancer immunotherapies potentially improve patient outcomes compared to results seen with single agents, in portions of the study to be added in the future, avelumab will be evaluated in combination with both standard-of-care chemotherapy and other anti-cancer immunotherapies in patients with advanced malignancies. Each cohort in the study will consist of a Phase 1b lead-in portion to evaluate safety and a Phase 2 cohort expansion to evaluate safety and efficacy.

In the Phase 1b safety lead-in portion, up to 12 patients will be enrolled into each cohort and evaluated for dose-limiting toxicities (DLT) during the first 2 cycles of treatment. If investigational products administration in a cohort is deemed safe in the Phase 1b lead-in, enrollment may be expanded into the Phase 2 cohort expansion. Up to approximately 40 patients in each cohort (including those enrolled in the Phase 1b lead-in and those enrolled in the Phase 2 cohort expansion) will be enrolled and treated with avelumab plus chemotherapy in the initial portion of the study and, in future portions of the study, with avelumab plus chemotherapy with or without other anti-cancer immunotherapies.

In the Phase 1b lead-in portions of NSCLC Cohort A1 and UC Cohort A2, avelumab is dosed at 800 mg fixed dose every 3 weeks. Under Protocol Amendment 4, avelumab is dosed at 1200 mg fixed dose every 3 weeks in the Phase 1b lead-in portions of NSCLC Cohort A3 and in UC Cohort A4, in combination with the same standard-of-care chemotherapy doublets used in Cohort A1 and Cohort A2, respectively. For each tumor type, the study treatment combination with the highest avelumab dose determined to be safe may be advanced into Phase 2 cohort expansion.

ELIGIBILITY:
Inclusion Criteria:

1. Histological diagnosis of locally advanced (primary or recurrent) or metastatic solid tumor that is not amenable for treatment with curative intent as follows:

   * For all groups:
   * Measurable disease by RECIST v1.1 with at least 1 measurable lesion, and availability of tumor specimen 18 months or less old.
   * No prior systemic treatment for unresectable locally advanced or metastatic disease for the tumor type under study. If prior systemic chemotherapy treatment was given in the adjuvant or neo-adjuvant setting or as part of radiotherapy chemotherapy treatment, disease-free interval after stop of systemic treatment must be more than 6 months for non-squamous NSCLC and more than 12 months for UC;
   * Cohort A1 and Cohort A3: Non-squamous NSCLC, with no activating EGFR mutations, ALK or ROS1 translocations/rearrangements. If monotherapy pembrolizumab is available as a standard of care treatment option, patients must have a tumor proportion score (TPS) <50% for PD L1 (via the 22C3 pharmDx or the Ventana (SP263) PD L1 IHC assay).
   * Cohort A2 and Cohort A4: Transitional cell carcinoma of the urothelium including the bladder, urethra, renal pelvis, and ureter.
2. ECOG performance status 0 or 1
3. Estimated life expectancy of at least 90 days
4. Adequate bone marrow, renal, and liver function
5. Negative serum pregnancy test at screening
6. Signed and dated informed consent

Exclusion Criteria:

1. Prior immunotherapy with any antibody or drug specifically targeting T cell co-stimulation or immune checkpoint pathways.
2. Patients with known symptomatic central nervous system metastases requiring steroids.
3. Diagnosis of other malignancy within 2 years prior to enrollment except adequately treated basal cell or squamous cell skin cancer, or carcinoma in situ of the bladder, breast, or cervix, or low grade (Gleason ≤6) prostate cancer
4. Use of immunosuppressive medication at the time of enrollment
5. Active or prior autoimmune disease that might deteriorate when receiving an immuno-stimulatory agent.
6. Prior organ transplantation including allogenic stem cell transplantation
7. Active infection requiring systemic therapy
8. Known history of HIV or AIDS
9. Hepatitis B virus (HBV) or hepatitis C virus (HCV) infection at screening
10. Administration of live vaccine within 4 weeks prior to study entry
11. Known prior severe hypersensitivity to the investigational products or any component in their formulations,
12. Known prior severe hypersensitivity to platinum-related compounds for all cohorts, to pemetrexed for patients enrolled in Cohort A1 and Cohort A3, and to gemcitabine for patients enrolled in Cohort A2 and Cohort A4
13. Persisting toxicity related to prior therapy (NCI CTCAE v4.03 Grade > 1)
14. Known history of colitis, inflammatory bowel disease, pneumonitis, pulmonary fibrosis.
15. Ongoing cardiac dysrhythmias of NCI CTCAE v4.03 Grade 2 or prolongation of the QTcF interval to >480 msec.
16. Clinically significant (ie, active) cardiovascular disease: cerebral vascular accident/stroke (<6 months prior to enrollment), myocardial infarction (< 6 months prior to enrollment), unstable angina, congestive heart failure, or serious cardiac arrhythmia requiring medication.
17. Major surgery ≤28 days or major radiation therapy ≤14 days prior to enrollment.
18. Participation in other studies involving investigational drug(s) within 28 days prior to study entry.
19. Concurrent treatment with a prohibited medication.
20. Other acute or chronic medical or psychiatric condition
21. Pregnant female patients; breastfeeding female patients; fertile male patients and female patients of childbearing potential who are unwilling or unable to use at least 1 highly effective method of contraception as outlined in this protocol for the duration of the study and for at least 90 days after the last dose of chemotherapy (for male and female patients) or at least 30 days after the last dose of avelumab (for female patients), whichever is longer.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2017-12-21 (Actual); Primary Completion 2021-06-07 (Actual); Study Completion 2022-12-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (40):
- United States (8):
  - University of Arizona Cancer Center - North Campus, Tucson, Arizona
  - Banner-University Medical Center Tucson, Tucson, Arizona
  - Stony Brook Cancer Center, Stony Brook, New York
  - Stony Brook University, Stony Brook, New York
  - Montefiore Medical Center - Einstein Center for Cancer Care, The Bronx, New York
  - Montefiore Medical Center - Moses Division, The Bronx, New York
  - Duke University Medical Center/Duke Cancer Center, Durham, North Carolina
  - Investigational Chemotherapy Service, Durham, North Carolina
- Australia (4):
  - Chris O'Brien Lifehouse, Camperdown, New South Wales
  - St Vincent's Hospital Sydney, Darlinghurst, New South Wales
  - St Vincent's Public Hospital Sydney, Darlinghurst, New South Wales
  - Western Health, Sunshine Hospital, St Albans, Victoria
- Kingston Health Sciences Centre -, Kingston, Ontario, Canada
- Czechia (6):
  - Fakultni nemocnice Olomouc, Klinika nuklearni mediciny, Olomouc
  - Fakultni nemocnice Olomouc, Ustav klinicke a molekularni patologie, Olomouc
  - Fakultni nemocnice Olomouc, Olomouc
  - Vseobecna fakultni nemocnice v Praze, Prague
  - Thomayerova nemocnice, Prague
  - Centrum nuklearni mediciny s.r.o., Prague
- Orszagos Onkologiai Intezet "C" Belgyogyaszati - Onkologiai es Klinikai Farmakologiai Osztaly, Budapest, Hungary
- Italy (6):
  - AOU Ospedali Riuniti di Ancona Umberto I - GM Lancisi - G Salesi, Torrette Di Ancona, AN
  - IRCCS Istit.Scient.Romagnolo per lo Studio e la Cura dei Tumori, Meldola, FC
  - Centro di Ricerca di Fase 1, ASST Monza-Ospedale San Gerardo, Monza, MB
  - Oncologia, ASST Monza-Ospedale San Gerardo, Monza, MB
  - Istituto Europeo di Oncologia (IEO), Milan, MI
  - Istituto Nazionale Tumori di Napoli IRCCS Fondazione Pascale, Napoli
- Spain (5):
  - Hospital Universitario Vall d'Hebron, Barcelona
  - Hospital Clinic I Provincial, Barcelona
  - Hospital Universitario Fundacion Jimenez Diaz, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Fundacion Instituto Valenciano de Oncologia, Valencia
- United Kingdom (9):
  - Royal Cornwall Hospital, Truro, Cornwall
  - The Platinum Medical Centre, London, England
  - The Wellington Hospital - South, London, England
  - Sarah Cannon Research Institute UK, London, England
  - The Harley Street Clinic, London, England
  - HCA Pharmacy Department, London, England
  - The Princess Grace Hospital, London, England
  - Weston Park Hospital, Sheffield, South Yorkshire
  - Sir Bobby Robson Cancer Trials Research Centre, Newcastle upon Tyne

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- [Derived] Wheatley DA, Berardi R, Climent Duran MA, Tomiak A, Greystoke AP, Joshua AM, Arkenau HT, Geczi L, Corbacho JG, Paz-Ares LG, Hussain SA, Petruzelka L, Delmonte A, Chappey C, Masters JC, Michelon E, Murphy DA, Mwewa S, Cesari R, Doger de Speville B. First-line Avelumab plus Chemotherapy in Patients with Advanced Solid Tumors: Results from the Phase Ib/II JAVELIN Chemotherapy Medley Study. Cancer Res Commun. 2024 Jun 28;4(6):1609-1619. doi: 10.1158/2767-9764.CRC-23-0459. PMID 38669053
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=B9991023

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted in 2 phases: Phase 1b (lead-in phase) and Phase 2 (cohort expansion phase). Phase 2 was conducted at the highest dose level of avelumab which was determined safe for participants in Phase 1b.
Pre-assignment Details: Phase 1b lead-in:49 participants signed inform consent form(ICF).18 participants did not meet eligibility criteria and not enrolled,31 participants enrolled and assigned to treatment. Phase 2:52 participants signed ICF.16 participants did not meet eligibility criteria and not enrolled,36 participants enrolled,1 was not assigned to treatment and 35 assigned to treatment.
Groups:
- Phase 1b Lead-in: Avelumab 800 mg + Pemetrexed/Carboplatin: Participants with advanced non-squamous non-small cell lung cancer (NSCLC) received avelumab 800 milligrams (mg) as an intravenous (IV) infusion over 1 hour every 3 weeks (Q3W) in combination with IV infusion of pemetrexed 500 milligram per square meter (mg/m^2) and carboplatin dose at area under curve (AUC) 5 (carboplatin dose [mg] = target AUC * glomerular filtration rate[GFR] milliliter per minute [mL/min] + 25, and maximum carboplatin dose = target AUC [mg*min/mL] * 150 mL/min) on Day 1 of each 21-day cycle. Pemetrexed/carboplatin were administered for a maximum of 4 to 6 cycles. Safety follow-up was for 90 days after last dose of study treatment or until time of initiation of new anticancer treatment, whichever comes first.
- Phase 1b Lead-in: Avelumab 800 mg + Gemcitabine/Cisplatin: Participants (cisplatin-eligible) with urothelial cancer (UC) received avelumab 800 mg as an IV infusion over 1 hour Q3W in combination with IV administration of cisplatin 70 mg/m^2 and gemcitabine 1000 mg/m^2 on Day 1 of each 21-day cycle with gemcitabine being administered on Day 1 and Day 8. Safety follow-up was for 90 days after last dose of study treatment or until time of initiation of new anticancer treatment, whichever comes first.
- Phase 1b Lead-in: Avelumab 1200 mg + Pemetrexed/Carboplatin: Participants with advanced NSCLC received avelumab 1200 mg as an IV infusion over 1 hour Q3W in combination with IV infusion of pemetrexed 500 mg/m^2 and carboplatin dose at AUC 5 (carboplatin dose [mg] = target AUC * GFR mL/min + 25), and maximum carboplatin dose = target AUC [mg*min/mL] * 150 mL/min) on Day 1 of each 21-day cycle. Pemetrexed/carboplatin were administered for a maximum of 4 to 6 cycles. Safety follow-up was for 90 days after last dose of study treatment or until time of initiation of new anticancer treatment, whichever comes first.
- Phase 1b Lead-in: Avelumab 1200 mg + Gemcitabine/Cisplatin; Phase 2: Avelumab 1200 mg + Gemcitabine/Cisplatin: Participants (cisplatin-eligible) with UC received avelumab 1200 mg as an IV infusion over 1 hour Q3W in combination with IV administration of cisplatin 70 mg/m^2 and gemcitabine 1000 mg/m^2 on Day 1 of each 21-day cycle with gemcitabine being administered on Day 1 and Day 8. Safety follow-up was for 90 days after last dose of study treatment or until time of initiation of new anticancer treatment, whichever comes first.
Period: Phase 1b Lead-in: Treatment
Arm/Group | Phase 1b Lead-in: Avelumab 800 mg + Pemetrexed/Carboplatin | Phase 1b Lead-in: Avelumab 800 mg + Gemcitabine/Cisplatin | Phase 1b Lead-in: Avelumab 1200 mg + Pemetrexed/Carboplatin | Phase 1b Lead-in: Avelumab 1200 mg + Gemcitabine/Cisplatin | Phase 2: Avelumab 1200 mg + Gemcitabine/Cisplatin
Started | 6 | 13 | 6 | 6 | 0
Completed | 0 | 0 | 0 | 0 | 0
Not Completed | 6 | 13 | 6 | 6 | 0
Not completed — Adverse Event | 3 | 4 | 1 | 1 | 0
Not completed — Physician Decision | 0 | 1 | 0 | 0 | 0
Not completed — Death | 0 | 0 | 1 | 0 | 0
Not completed — Progressive Disease | 1 | 6 | 3 | 4 | 0
Not completed — Other | 2 | 1 | 0 | 0 | 0
Not completed — Global deterioration of health status | 0 | 0 | 1 | 0 | 0
Not completed — Study terminated by sponsor | 0 | 1 | 0 | 1 | 0
Period: Phase 1b Lead-in: Follow-up
Arm/Group | Phase 1b Lead-in: Avelumab 800 mg + Pemetrexed/Carboplatin | Phase 1b Lead-in: Avelumab 800 mg + Gemcitabine/Cisplatin | Phase 1b Lead-in: Avelumab 1200 mg + Pemetrexed/Carboplatin | Phase 1b Lead-in: Avelumab 1200 mg + Gemcitabine/Cisplatin | Phase 2: Avelumab 1200 mg + Gemcitabine/Cisplatin
Started | 6 (Eligible participants entered follow-up period following discontinuation of study treatment) | 12 (Eligible participants entered follow-up period following discontinuation of study treatment) | 5 (Eligible participants entered follow-up period following discontinuation of study treatment) | 6 (Eligible participants entered follow-up period following discontinuation of study treatment) | 0
Completed | 0 | 0 | 0 | 0 | 0
Not Completed | 6 | 12 | 5 | 6 | 0
Not completed — Death | 3 | 8 | 4 | 4 | 0
Not completed — Lost to Follow-up | 1 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 0 | 0
Not completed — Other | 0 | 1 | 0 | 1 | 0
Not completed — Study terminated by sponsor | 2 | 3 | 0 | 1 | 0
Period: Phase 2: Treatment
Arm/Group | Phase 1b Lead-in: Avelumab 800 mg + Pemetrexed/Carboplatin | Phase 1b Lead-in: Avelumab 800 mg + Gemcitabine/Cisplatin | Phase 1b Lead-in: Avelumab 1200 mg + Pemetrexed/Carboplatin | Phase 1b Lead-in: Avelumab 1200 mg + Gemcitabine/Cisplatin | Phase 2: Avelumab 1200 mg + Gemcitabine/Cisplatin
Started | 0 | 0 | 0 | 0 | 35 (Additional participants were enrolled in Phase 2)
Completed | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 35
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 6
Not completed — Progressive disease | 0 | 0 | 0 | 0 | 22
Not completed — Other | 0 | 0 | 0 | 0 | 4
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 1
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 1
Not completed — Death | 0 | 0 | 0 | 0 | 1
Period: Phase 2: Follow-up
Arm/Group | Phase 1b Lead-in: Avelumab 800 mg + Pemetrexed/Carboplatin | Phase 1b Lead-in: Avelumab 800 mg + Gemcitabine/Cisplatin | Phase 1b Lead-in: Avelumab 1200 mg + Pemetrexed/Carboplatin | Phase 1b Lead-in: Avelumab 1200 mg + Gemcitabine/Cisplatin | Phase 2: Avelumab 1200 mg + Gemcitabine/Cisplatin
Started | 0 | 0 | 0 | 0 | 33 (Eligible participants entered follow-up period following discontinuation of study treatment)
Completed | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 33
Not completed — Death | 0 | 0 | 0 | 0 | 24
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 1
Not completed — Other | 0 | 0 | 0 | 0 | 1
Not completed — Study terminated by sponsor | 0 | 0 | 0 | 0 | 7

BASELINE CHARACTERISTICS:
Groups:
- Phase 1b Lead-in+Phase 2:Avelumab 1200mg+Gemcitabine/Cisplatin: Participants (cisplatin-eligible) with UC received avelumab 1200 mg as an IV infusion over 1 hour Q3W in combination with IV administration of cisplatin 70 mg/m^2 and gemcitabine 1000 mg/m^2 on Day 1 of each 21-day cycle with gemcitabine being administered on Day 1 and Day 8. Safety follow-up was for 90 days after last dose of study treatment or until time of initiation of new anticancer treatment, whichever comes first. Participants from both Phase 1b and Phase 2 Avelumab 1200 mg + Gemcitabine/Cisplatin were included in this arm.
- Total: Total of all reporting groups
Arm/Group | Phase 1b Lead-in: Avelumab 800 mg + Pemetrexed/Carboplatin | Phase 1b Lead-in: Avelumab 800 mg + Gemcitabine/Cisplatin | Phase 1b Lead-in: Avelumab 1200 mg + Pemetrexed/Carboplatin | Phase 1b Lead-in+Phase 2:Avelumab 1200mg+Gemcitabine/Cisplatin | Total
Number analyzed (Participants) | 6 | 13 | 6 | 41 | 66
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 1 | 7 | 3 | 14 | 25
  >=65 years | 5 | 6 | 3 | 27 | 41
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 5 | 0 | 10 | 17
  Male | 4 | 8 | 6 | 31 | 49
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 0 | 0 | 1
  Not Hispanic or Latino | 6 | 11 | 6 | 37 | 60
  Unknown or Not Reported | 0 | 1 | 0 | 4 | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 1 | 1 | 1 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 1 | 0 | 0 | 1
  White | 6 | 11 | 5 | 37 | 59
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 3 | 3

OUTCOME MEASURES:

1. Secondary Outcome: Serum Concentration of Avelumab
Description: The lower limit of quantification (LLOQ) for avelumab was 0.2 micrograms per milliliter. Pharmacokinetic concentration analysis set was subset of safety analysis set and included participants who had at least one concentration measurement for avelumab or other study drugs which they were assigned to receive. Treatment groups with same dose and administration frequency were combined as pre-specified in reporting and analysis plan.
Time Frame: Pre-dose, 1 hour post-dose on Day 1 of Cycle 1, 2, 3, 6, 10, 14; 336 hours post-dose on Day 15 of Cycle 1, 2, 3 (each cycle of 21 days)
Population: The PK concentration analysis sets are subsets of the safety analysis set including participants who have at least one concentration measurement for avelumab which they were assigned to receive,based on the treatment group.Overall number of participants analyzed=participants evaluable for this outcome measure and only those contributing to data for this outcome measure.Number analyzed=participants evaluable and contributing at specified time point.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Micrograms per milliliter
Arm/Group | Phase 1b Lead-in: Avelumab 800 mg + Pemetrexed/Carboplatin | Phase 1b Lead-in: Avelumab 800 mg + Gemcitabine/Cisplatin | Phase 1b Lead-in: Avelumab 1200 mg + Pemetrexed/Carboplatin | Phase 1b Lead-in+Phase 2:Avelumab 1200mg+Gemcitabine/Cisplatin
Number analyzed (Participants) | 6 | 13 | 6 | 40
Micrograms per milliliter
  Cycle 1/Day 1- 1 hour: number analyzed (Participants) | 4 | 10 | 4 | 32
  Cycle 1/Day 1- 1 hour | 173.3 (26) | 172.2 (18) | 284.1 (33) | 300.2 (32)
  Cycle 1/Day 15- 336 hours: number analyzed (Participants) | 6 | 12 | 6 | 34
  Cycle 1/Day 15- 336 hours | 12.32 (47) | 9.570 (92) | 16.51 (68) | 14.71 (74)
  Cycle 2/Day 1- pre-dose: number analyzed (Participants) | 6 | 8 | 6 | 24
  Cycle 2/Day 1- pre-dose | 4.780 (44) | 3.754 (115) | 4.328 (332) | 5.013 (196)
  Cycle 2/Day 1- 1 hour: number analyzed (Participants) | 4 | 8 | 4 | 20
  Cycle 2/Day 1- 1 hour | 164.2 (33) | 197.0 (18) | 104.5 (1474) | 311.9 (36)
  Cycle 2/Day 15- 336 hours: number analyzed (Participants) | 6 | 8 | 5 | 27
  Cycle 2/Day 15- 336 hours | 16.87 (24) | 13.55 (33) | 16.82 (137) | 18.66 (75)
  Cycle 3/Day 1- pre-dose: number analyzed (Participants) | 5 | 9 | 5 | 19
  Cycle 3/Day 1- pre-dose | 8.122 (40) | 5.651 (75) | 4.878 (662) | 6.771 (104)
  Cycle 3/Day 1- 1 hour: number analyzed (Participants) | 4 | 7 | 4 | 11
  Cycle 3/Day 1- 1 hour | 147.0 (35) | 204.0 (28) | 93.81 (2989) | 296.8 (36)
  Cycle 3/Day 15- 336 hours: number analyzed (Participants) | 5 | 7 | 6 | 16
  Cycle 3/Day 15- 336 hours | 19.40 (14) | 17.15 (40) | 26.17 (74) | 22.55 (79)
  Cycle 6/Day 1- pre-dose: number analyzed (Participants) | 5 | 7 | 4 | 19
  Cycle 6/Day 1- pre-dose | 11.38 (24) | 9.518 (65) | 10.86 (165) | 10.39 (233)
  Cycle 6/Day 1- 1 hour: number analyzed (Participants) | 4 | 7 | 3 | 12
  Cycle 6/Day 1- 1 hour | 92.53 (203) | 208.3 (23) | 245.4 (6) | 344.0 (27)
  Cycle 10/Day 1- pre-dose: number analyzed (Participants) | 4 | 6 | 1 | 14
  Cycle 10/Day 1- pre-dose | 9.523 (33) | 8.695 (115) | 6.620 (NA) — Data was not estimable due to low number of participants analyzed. | 18.55 (58)
  Cycle 10/Day 1- 1 hour: number analyzed (Participants) | 3 | 6 | 1 | 6
  Cycle 10/Day 1- 1 hour | 179.0 (38) | 222.0 (27) | 6.040 (NA) — Data was not estimable due to low number of participants analyzed. | 242.9 (121)
  Cycle 14/Day 1- pre-dose: number analyzed (Participants) | 3 | 4 | 2 | 8
  Cycle 14/Day 1- pre-dose | 14.97 (28) | 13.37 (77) | 12.24 (523) | 16.49 (57)
  Cycle 14/Day 1- 1 hour: number analyzed (Participants) | 3 | 4 | 2 | 5
  Cycle 14/Day 1- 1 hour | 215.3 (20) | 216.6 (22) | 29.05 (20555) | 402.2 (19)

2. Secondary Outcome: Absolute Value of Tumor Mutational Burden (TMB) in Tumor Tissue
Description: Mutational load within tumor tissue was defined as number per megabase of the genome, coding, base substitution, and indel mutations present in the sample. Mutational load was determined in whole blood samples using next generation deoxyribonucleic acid (DNA) sequencing followed by computational analysis.
Time Frame: Pre-dose on Day 1 of Cycle 1
Population: The tumor tissue-based biomarker analysis set was subset of the safety analysis set and included participants who had at least one baseline and one on-treatment biomarker assessment for the same biomarker. Treatment groups with same dose and administration frequency were combined as pre-specified in reporting and analysis plan.
Measure: Mean (Standard Deviation); unit: Mutations per megabase
Arm/Group | Phase 1b Lead-in: Avelumab 800 mg + Pemetrexed/Carboplatin | Phase 1b Lead-in: Avelumab 800 mg + Gemcitabine/Cisplatin | Phase 1b Lead-in: Avelumab 1200 mg + Pemetrexed/Carboplatin | Phase 1b Lead-in+Phase 2:Avelumab 1200mg+Gemcitabine/Cisplatin
Number analyzed (Participants) | 4 | 13 | 5 | 39
Mutations per megabase | 4.3 (6.75) [lower limit 6.75] | 2.8 (2.76) [lower limit 2.76] | 4.4 (5.15) [lower limit 5.15] | 2.5 (2.88) [lower limit 2.88]

3. Primary Outcome: Phase 1b Lead-in: Number of Participants With Dose-Limiting Toxicities (DLT)
Description: DLTs=occurrence of any AEs attributable to study treatment in first 2 treatment cycles:Hematologic: grade(G)4 neutropenia lasting >7days;febrile neutropenia with body temperature >=38 degree Celsius for >1hour; G>=3 neutropenic infection(absolute neutrophil count <1.0*10^9/L),G>=3 thrombocytopenia (platelet count<50.0-25.0*10^9/L)with bleeding;G4 thrombocytopenia(PC<25.0*10^9/L),G4 anemia(life-threatening).Non-hematologic: any G4 toxicities;G3 toxicities persisting for >3days despite medical treatment(nausea,vomiting,diarrhea)except endocrinopathies controlled with hormonal therapy;ALT/AST >3*upper limit of normal(ULN)if normal at baseline or 2*Baseline(>ULN at baseline)with total bilirubin >2*ULN and alkaline phosphatase <2*ULN;G3 QTcF prolongation after correction of any reversible cause(electrolyte abnormalities/hypoxia).Delay of >=3weeks in scheduled administration/failure to deliver 75% of doses due to toxicities attributable to any study treatment. DLT-evaluable analysis set.
Time Frame: Day 1 up to Week 6 (first 2 treatment cycles; 1 cycle = 21 days)
Population: The DLT analysis set is a subset of the safety analysis set and includes all enrolled participants in the Phase 1b lead-in who are eligible for the study, receive at least one dose of the combination treatment, and either experience DLT during the first 2 cycles (6 weeks) of treatment, or complete the DLT observation period for the first 2 cycles of treatment.
Measure: Count of Participants; unit: Participants
Groups:
- Phase 1b Lead-in: Avelumab 1200mg+Gemcitabine/Cisplatin: Participants (cisplatin-eligible) with UC received avelumab 1200 mg as an IV infusion over 1 hour Q3W in combination with IV administration of cisplatin 70 mg/m^2 and gemcitabine 1000 mg/m^2 on Day 1 of each 21-day cycle with gemcitabine being administered on Day 1 and Day 8. Safety follow-up was for 90 days after last dose of study treatment or until time of initiation of new anticancer treatment, whichever comes first.
Arm/Group | Phase 1b Lead-in: Avelumab 800 mg + Pemetrexed/Carboplatin | Phase 1b Lead-in: Avelumab 800 mg + Gemcitabine/Cisplatin | Phase 1b Lead-in: Avelumab 1200 mg + Pemetrexed/Carboplatin | Phase 1b Lead-in: Avelumab 1200mg+Gemcitabine/Cisplatin
Number analyzed (Participants) | 6 | 12 | 6 | 6
Participants | 0 | 1 | 0 | 1

4. Primary Outcome: Percentage of Participants With Confirmed Objective Response (OR) as Per Response Evaluation Criteria in Solid Tumors (RECIST) Version (v) 1.1 by Investigator Assessment
Description: OR: complete response(CR) or partial response(PR)determined by investigator according to RECIST v1.1 from date of first dose of study treatment until date of first documentation of progressive disease(PD),confirmed by repeat assessments performed no less than 4 weeks after first response. CR: disappearance of target and non-target lesions, with exception of nodal disease and normalization of tumor markers. All nodes, target and non-target must have short axis measures less than (<)10 millimeter(mm). PR: >=30% decrease in sum of measures (longest diameter for tumor lesions and short axis measure for nodes) of target lesions, taking as reference baseline sum of diameters. Non-target lesions must be non-PD. PD: >=20% increase in sum of diameters of target lesions, taking as reference the smallest sum on study. In addition to relative increase of 20%, sum must also demonstrate an absolute increase of at least 5mm, appearance of one or more new lesions was considered PD.
Time Frame: From start of the treatment until disease progression or death due to any cause, whichever occurred first (maximum up to 3.5 years approximately)
Population: The full analysis set (FAS) will include all participants who receive at least one dose of study drug. Participants will be classified according to the study treatment actually received. If a participant receives more than one treatment the participant will be classified according to the first study treatment received.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Phase 1b Lead-in: Avelumab 800 mg + Pemetrexed/Carboplatin | Phase 1b Lead-in: Avelumab 800 mg + Gemcitabine/Cisplatin | Phase 1b Lead-in: Avelumab 1200 mg + Pemetrexed/Carboplatin | Phase 1b Lead-in+Phase 2:Avelumab 1200mg+Gemcitabine/Cisplatin
Number analyzed (Participants) | 6 | 13 | 6 | 41
Percentage of Participants | 50.0 (11.8) [11.8 to 88.2] | 53.8 (25.1) [25.1 to 80.8] | 33.3 (4.3) [4.3 to 77.7] | 39.0 (24.2) [24.2 to 55.5]

5. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs) and Serious TEAEs
Description: Adverse event (AE) was any untoward medical occurrence in a participants who received any study drug without regard to possibility of causal relationship. Serious adverse event was any untoward medical occurrence that at any dose resulted in any of following outcomes/deemed significant for any other reason: death; initial /prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly/birth defect. TEAEs were those events with onset dates occurring during the on-treatment period. On-treatment period was defined as time from first dose of any study treatment and up to 30 days after last dose or start day of new anti-cancer drug therapy minus 1 day, whichever occurred first.
Time Frame: From start of the treatment up to 30 days after last dose or start of new anticancer therapy minus 1 day, whichever occurred first (maximum up to 5 years approximately)
Population: Safety analysis set included all participants who received at least 1 dose of any study drug. Treatment groups with same dose and administration frequency were combined as pre-specified in reporting and analysis plan.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1b Lead-in: Avelumab 800 mg + Pemetrexed/Carboplatin | Phase 1b Lead-in: Avelumab 800 mg + Gemcitabine/Cisplatin | Phase 1b Lead-in: Avelumab 1200 mg + Pemetrexed/Carboplatin | Phase 1b Lead-in+Phase 2:Avelumab 1200mg+Gemcitabine/Cisplatin
Number analyzed (Participants) | 6 | 13 | 6 | 41
Participants
  TEAEs | 6 | 13 | 6 | 40
  Serious TEAEs | 3 | 9 | 5 | 20

6. Secondary Outcome: Number of Participants With Treatment Related TEAEs
Description: A treatment related AE included AEs related to at least one study drug in the combination. TEAEs were those events with onset dates occurring during the on-treatment period. On-treatment period was defined as time from first dose of any study treatment and up to 30 days after last dose or start day of new anti-cancer drug therapy minus 1 day, whichever occurred first. Relatedness to study drug was assessed by the investigator.
Time Frame: as for outcome 5
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1b Lead-in: Avelumab 800 mg + Pemetrexed/Carboplatin | Phase 1b Lead-in: Avelumab 800 mg + Gemcitabine/Cisplatin | Phase 1b Lead-in: Avelumab 1200 mg + Pemetrexed/Carboplatin | Phase 1b Lead-in+Phase 2:Avelumab 1200mg+Gemcitabine/Cisplatin
Number analyzed (Participants) | 6 | 13 | 6 | 41
Participants | 6 | 12 | 6 | 40

7. Secondary Outcome: Number of Participants With Grade 3 or Higher TEAEs Based on National Cancer Institute Common Toxicity Criteria for Adverse Events (NCI CTCAE) v 4.03
Description: AE was any untoward medical occurrence in a participant who received any study drug without regard to possibility of causal relationship. TEAEs were those events with onset dates occurring during the on-treatment period. On-treatment period was defined as time from first dose of any study treatment and up to 30 days after last dose or start day of new anti-cancer drug therapy minus 1 day, whichever occurred first. TEAEs were graded by the investigator using NCI CTCAE v 4.03 as Grade 1 = mild; Grade 2 = moderate; Grade 3 = severe; Grade 4 = life-threatening; Grade 5 = death. In this outcome measure, number of participants with grade 3 or higher TEAEs were reported.
Time Frame: as for outcome 5
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1b Lead-in: Avelumab 800 mg + Pemetrexed/Carboplatin | Phase 1b Lead-in: Avelumab 800 mg + Gemcitabine/Cisplatin | Phase 1b Lead-in: Avelumab 1200 mg + Pemetrexed/Carboplatin | Phase 1b Lead-in+Phase 2:Avelumab 1200mg+Gemcitabine/Cisplatin
Number analyzed (Participants) | 6 | 13 | 6 | 41
Participants | 5 | 12 | 6 | 37

8. Secondary Outcome: Number of Participants With Grade 3 or Higher Laboratory Abnormalities by CTCAE Grade
Description: Participants with laboratory abnormalities of any Grade as per NCI CTCAE toxicity grading v4.03 were summarized:hematology(anemia,hemoglobin increased,lymphocyte count decreased,lymphocyte count increased, neutrophil count decreased,platelet count decreased and white blood cell decreased)and clinical chemistry(alanine aminotransferase increased,alkaline phosphatase,increased,aspartate,aminotransferase increased,blood bilirubin increased,cholesterol high,creatinine phosphokinase[cpk] increased,creatinine increased,gamma-glutamyl transferase[ggt] increased,hypercalcemia,hyperglycemia,hyperkalemia, hypermagnesemia,hypernatremia,hypertriglyceridemia,hypoalbuminemia,hypocalcemia,hypoglycemia,hypokalemia,hypomagnesemia,hyponatremia, hypophosphatemia,serum amylase increased and lipase increased).As per NCI CTCAE toxicity grading v4.03, Grade1=mild;Grade2=moderate;Grade3=severe;Grade4=life-threatening;Grade 5=death.Parameters with at least 1 participant with abnormal value are reported.
Time Frame: From screening up to 90 days after last dose of study drug (maximum up to 5 years approximately)
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1b Lead-in: Avelumab 800 mg + Pemetrexed/Carboplatin | Phase 1b Lead-in: Avelumab 800 mg + Gemcitabine/Cisplatin | Phase 1b Lead-in: Avelumab 1200 mg + Pemetrexed/Carboplatin | Phase 1b Lead-in+Phase 2:Avelumab 1200mg+Gemcitabine/Cisplatin
Number analyzed (Participants) | 6 | 13 | 6 | 40
Participants
  ALANINE AMINOTRANSFERASE INCREASED | 1 | 1 | 0 | 3
  ALKALINE PHOSPHATASE INCREASED | 0 | 0 | 0 | 1
  ASPARTATE AMINOTRANSFERASE INCREASED | 1 | 1 | 0 | 2
  BLOOD BILIRUBIN INCREASED | 0 | 1 | 0 | 0
  CPK INCREASED | 0 | 0 | 0 | 1
  CREATININE INCREASED | 1 | 1 | 0 | 0
  GGT INCREASED | 0 | 2 | 1 | 4
  HYPERGLYCEMIA | 2 | 2 | 0 | 4
  HYPERKALEMIA | 0 | 1 | 0 | 2
  HYPOKALEMIA | 1 | 0 | 0 | 5
  HYPONATREMIA | 0 | 2 | 1 | 4
  LIPASE INCREASED | 1 | 2 | 1 | 4
  SERUM AMYLASE INCREASED | 0 | 2 | 0 | 4
  HYPOPHOSPHATEMIA | 2 | 0 | 1 | 3
  HYPOMAGNESEMIA | 0 | 0 | 0 | 2
  HYPOCALCEMIA | 2 | 0 | 0 | 1
  HYPERTRIGLYCERIDEMIA | 0 | 3 | 0 | 2
  HYPERNATREMIA | 0 | 0 | 0 | 1
  HYPERMAGNESEMIA | 0 | 0 | 0 | 1
  HYPERCALCEMIA | 0 | 0 | 0 | 1
  ANEMIA | 2 | 5 | 0 | 6
  LYMPHOCYTE COUNT DECREASED | 3 | 5 | 1 | 7
  LYMPHOCYTE COUNT INCREASED | 0 | 0 | 0 | 1
  NEUTROPHIL COUNT DECREASED | 3 | 8 | 3 | 21
  PLATELET COUNT DECREASED | 3 | 2 | 0 | 11
  WHITE BLOOD CELL DECREASED | 2 | 7 | 3 | 16

9. Secondary Outcome: Number of Participants With Positive Anti-Drug Antibody (ADA) and Neutralizing Antibodies for Avelumab
Description: Blood samples were collected for assessment of avelumab ADAs using a tiered assay and confirmed positive samples were tested for neutralizing antibodies (nAb).
Time Frame: From first dose of study drug up to last dose of study drug (maximum up to 5 years approximately)
Population: The immunogenicity analysis set is a subset of the safety analysis set and will include participants who have at least one ADA/nAb sample collected for avelumab.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1b Lead-in: Avelumab 800 mg + Pemetrexed/Carboplatin | Phase 1b Lead-in: Avelumab 800 mg + Gemcitabine/Cisplatin | Phase 1b Lead-in: Avelumab 1200 mg + Pemetrexed/Carboplatin | Phase 1b Lead-in+Phase 2:Avelumab 1200mg+Gemcitabine/Cisplatin
Number analyzed (Participants) | 6 | 13 | 6 | 41
Participants
  ADA ever positive | 0 | 5 | 1 | 9
  NAB ever positive | NA — The data for NAB was not generated due to low observed immunogenicity. | NA — The data for NAB was not generated due to low observed immunogenicity. | NA — The data for NAB was not generated due to low observed immunogenicity. | NA — The data for NAB was not generated due to low observed immunogenicity.

10. Secondary Outcome: Progression Free Survival (PFS) as Per RECIST v 1.1 by Investigator Assessment
Description: PFS was defined as the time from the date of first dose of study treatment to the date of the first documentation of PD per RECIST v1.1 or death due to any cause, whichever occurred first. PD: >=20% increase in sum of diameters of target lesions, taking as reference the smallest sum on study. In addition to relative increase of 20%, sum must also demonstrate an absolute increase of at least 5mm, appearance of one or more new lesions was considered PD. The median duration of PFS was not derived for less than (<) 10 participants.
Time Frame: From start of treatment until disease progression or death due to any cause, whichever occurred first (maximum up to 5 years approximately)
Population: The full analysis set (FAS) included all participants who received at least 1 dose of study drug. Treatment groups with same dose and administration frequency were combined as pre-specified in reporting and analysis plan.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Phase 1b Lead-in: Avelumab 800 mg + Pemetrexed/Carboplatin | Phase 1b Lead-in: Avelumab 800 mg + Gemcitabine/Cisplatin | Phase 1b Lead-in: Avelumab 1200 mg + Pemetrexed/Carboplatin | Phase 1b Lead-in+Phase 2:Avelumab 1200mg+Gemcitabine/Cisplatin
Number analyzed (Participants) | 6 | 13 | 6 | 41
Months | NA [NA to NA] — Median and 95% CI were not estimated for <10 participants. | 9.8 [2.2 to NA] — Upper limit of 95% CI was not reached due to fewer number of participants with event. | NA [NA to NA] — Median and 95% CI were not estimated for <10 participants. | 5.4 [2.9 to 6.0]

11. Secondary Outcome: Overall Survival (OS)
Description: OS was defined as the time from the first dose of study treatment to the date of death due to any cause. Participants last known to be alive were censored at the date of last contact. The median duration of OS was not derived for less than (<) 10 participants.
Time Frame: From first dose of study treatment until death due to any cause (maximum up to 5 years approximately)
Population: as for outcome 10
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Phase 1b Lead-in: Avelumab 800 mg + Pemetrexed/Carboplatin | Phase 1b Lead-in: Avelumab 800 mg + Gemcitabine/Cisplatin | Phase 1b Lead-in: Avelumab 1200 mg + Pemetrexed/Carboplatin | Phase 1b Lead-in+Phase 2:Avelumab 1200mg+Gemcitabine/Cisplatin
Number analyzed (Participants) | 6 | 13 | 6 | 41
Months | NA [NA to NA] — Median and 95% CI were not estimated for <10 participants. | 18.1 [5.0 to NA] — Upper limit of 95% CI was not reached due to fewer number of participants with event. | NA [NA to NA] — Median and 95% CI were not estimated for <10 participants. | 15.1 [8.7 to 22.0]

12. Secondary Outcome: Duration of Response (DOR) as Per RECIST v 1.1 by Investigator Assessment
Description: DOR was defined as time from first documentation of objective response (confirmed CR or PR) to the date of first PD documentation or death due to any cause, whichever occurs first. CR: disappearance of target and non-target lesions, with exception of nodal disease and normalization of tumor markers. All nodes, target and non-target must have short axis measures less than (<)10 millimeter(mm). PR: >=30% decrease in sum of measures (longest diameter for tumor lesions and short axis measure for nodes) of target lesions, taking as reference baseline sum of diameters. Non-target lesions must be non-PD. PD: >=20% increase in sum of diameters of target lesions, taking as reference the smallest sum on study. In addition to relative increase of 20%, sum must also demonstrate an absolute increase of at least 5mm, appearance of one or more new lesions was considered PD. Median DOR was not derived for < 5 participants.
Time Frame: From date of first documented response to date of first documented PD or death due to any cause, whichever occurred first (maximum up to 5 years approximately)
Population: as for outcome 10
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Phase 1b Lead-in: Avelumab 800 mg + Pemetrexed/Carboplatin | Phase 1b Lead-in: Avelumab 800 mg + Gemcitabine/Cisplatin | Phase 1b Lead-in: Avelumab 1200 mg + Pemetrexed/Carboplatin | Phase 1b Lead-in+Phase 2:Avelumab 1200mg+Gemcitabine/Cisplatin
Number analyzed (Participants) | 3 | 7 | 2 | 16
Months | NA [NA to NA] — Median and 95% CI were not estimated for <5 participants. | 9.6 [4.0 to NA] — Upper limit of 95% CI was not reached due to fewer number of participants with event. | NA [NA to NA] — Median and 95% CI were not estimated for <5 participants. | NA [4.2 to NA] — Median and Upper limit of 95% CI were not reached due to fewer number of participants with event.

13. Secondary Outcome: Time-to-Tumor Response (TTR) as Per RECIST v 1.1 by Investigator Assessment
Description: TTR was defined as the time from the date of first dose of study treatment to the first documentation of objective response (CR or PR) as assessed by investigator according to RECIST v 1.1. CR: disappearance of target and non-target lesions, with exception of nodal disease and normalization of tumor markers. All nodes, target and non-target must have short axis measures less than (<)10 millimeter(mm). PR: >=30% decrease in sum of measures (longest diameter for tumor lesions and short axis measure for nodes) of target lesions, taking as reference baseline sum of diameters. Non-target lesions must be non-PD.
Time Frame: From first dose of study treatment until first documentation of CR or PR (maximum up to 5 years approximately)
Population: as for outcome 10
Measure: Median (Full Range); unit: Months
Arm/Group | Phase 1b Lead-in: Avelumab 800 mg + Pemetrexed/Carboplatin | Phase 1b Lead-in: Avelumab 800 mg + Gemcitabine/Cisplatin | Phase 1b Lead-in: Avelumab 1200 mg + Pemetrexed/Carboplatin | Phase 1b Lead-in+Phase 2:Avelumab 1200mg+Gemcitabine/Cisplatin
Number analyzed (Participants) | 3 | 7 | 2 | 16
Months | 2.8 (1.3) [1.3 to 4.1] | 1.4 (1.1) [1.1 to 1.5] | 1.3 (1.3) [1.3 to 1.3] | 1.5 (1.3) [1.3 to 4.3]

14. Secondary Outcome: Number of Participants With Programmed Death-Ligand 1 (PD-L1) Expression
Description: PD-L1 expression was determined using the Ventana PD-L1 SP263 IHC assay. PD-L1-positive status in UC cohorts was defined using an algorithm that combines assessments of PD-L1 staining on tumor and immune cells scored by pathologists and in NSCLC cohorts was defined as PD-L1 expression on >=1% of tumor cells. PD-L1 expression at baseline and on-treatment were reported in this outcome measure.
Time Frame: Baseline and Cycle 2 Day 8 (each cycle of 21 days)
Population: FAS included all participants who received at least one dose of study drug. Treatment groups with same dose and administration frequency were combined as pre-specified in reporting and analysis plan.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1b Lead-in: Avelumab 800 mg + Pemetrexed/Carboplatin | Phase 1b Lead-in: Avelumab 800 mg + Gemcitabine/Cisplatin | Phase 1b Lead-in: Avelumab 1200 mg + Pemetrexed/Carboplatin | Phase 1b Lead-in+Phase 2:Avelumab 1200mg+Gemcitabine/Cisplatin
Number analyzed (Participants) | 6 | 13 | 6 | 41
Participants
  Baseline- Positive PD-L1 | 0 | 6 | 1 | 28
  Baseline- Negative PD-L1 | 4 | 7 | 4 | 13
  Baseline- Unknown PD-L1 | 2 | 0 | 1 | 0
  On-treatment (Cycle 2 Day 8)- Positive PD-L1 | 0 | 2 | 1 | 3
  On-treatment (Cycle 2 Day 8)- Negative PD-L1 | 2 | 1 | 0 | 6
  On-treatment (Cycle 2 Day 8)- Unknown PD-L1 | 4 | 10 | 5 | 32

ADVERSE EVENTS:
Time Frame: All-cause mortality: From start of the treatment up to 90 days post last dose of study treatment (maximum of 5 years approximately), TEAEs and Serious TEAEs: From start of the treatment up to 30 days post last dose of study treatment
Description: Same event may appear as both an AE and SAE. Safety set was evaluated. Treatment groups with same dose and administration frequency were combined as pre-specified in reporting and analysis plan.
Groups:
- Phase 1b and 2: Avelumab 1200 mg + Gemcitabine/Cisplatin: Participants (cisplatin-eligible) with UC received avelumab 1200 mg as an IV infusion over 1 hour Q3W in combination with IV administration of cisplatin 70 mg/m^2 and gemcitabine 1000 mg/m^2 on Day 1 of each 21-day cycle with gemcitabine being administered on Day 1 and Day 8. Safety follow-up was for 90 days after last dose of study treatment or until time of initiation of new anticancer treatment, whichever comes first. Participants from both Phase 1b and Phase 2 Avelumab 1200 mg + Gemcitabine/Cisplatin were included in this arm.
Arm/Group | Phase 1b Lead-in: Avelumab 800 mg + Pemetrexed/Carboplatin | Phase 1b Lead-in: Avelumab 800 mg + Gemcitabine/Cisplatin | Phase 1b Lead-in: Avelumab 1200 mg + Pemetrexed/Carboplatin | Phase 1b and 2: Avelumab 1200 mg + Gemcitabine/Cisplatin
All-Cause Mortality (participants affected / at risk) | 3/6 | 8/13 | 5/6 | 29/41
Serious Adverse Events (participants affected / at risk) | 3/6 | 9/13 | 5/6 | 20/41
Other Adverse Events (participants affected / at risk) | 6/6 | 13/13 | 6/6 | 40/41
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phase 1b Lead-in: Avelumab 800 mg + Pemetrexed/Carboplatin (N=6) | Phase 1b Lead-in: Avelumab 800 mg + Gemcitabine/Cisplatin (N=13) | Phase 1b Lead-in: Avelumab 1200 mg + Pemetrexed/Carboplatin (N=6) | Phase 1b and 2: Avelumab 1200 mg + Gemcitabine/Cisplatin (N=41)
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
Pancytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1
Atrial thrombosis (Cardiac disorders) | 0 | 1 | 0 | 0
Atrioventricular block (Cardiac disorders) | 0 | 1 | 0 | 0
Bradycardia (Cardiac disorders) | 0 | 0 | 0 | 1
Cardiomyopathy (Cardiac disorders) | 0 | 0 | 0 | 1
Myocardial infarction (Cardiac disorders) | 0 | 2 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Colitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 1 | 0 | 0
Ileus (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Pancreatitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Subileus (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Autoimmune hepatitis (Hepatobiliary disorders) | 0 | 0 | 0 | 1
Bacteraemia (Infections and infestations) | 0 | 0 | 0 | 1
Bacteriuria (Infections and infestations) | 0 | 0 | 0 | 1
Infection (Infections and infestations) | 0 | 0 | 0 | 1
Pyelonephritis (Infections and infestations) | 0 | 0 | 0 | 1
Rectal abscess (Infections and infestations) | 0 | 0 | 1 | 0
Rhinovirus infection (Infections and infestations) | 0 | 1 | 0 | 0
Sepsis (Infections and infestations) | 0 | 1 | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 2 | 0 | 5
Urosepsis (Infections and infestations) | 0 | 1 | 0 | 0
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 2
Spinal fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 0 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Fasciitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 0 | 1 | 0 | 0
Hydrocephalus (Nervous system disorders) | 0 | 0 | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 1 | 1 | 0 | 0
Renal impairment (Renal and urinary disorders) | 0 | 0 | 0 | 1
Urinary retention (Renal and urinary disorders) | 0 | 1 | 0 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1
Hypotension (Vascular disorders) | 0 | 1 | 0 | 0
Peripheral embolism (Vascular disorders) | 0 | 1 | 0 | 0
Malaise (General disorders) | 0 | 0 | 0 | 1
Sudden death (General disorders) | 0 | 0 | 0 | 1
Haematuria (Renal and urinary disorders) | 0 | 0 | 0 | 1
Renal haemorrhage (Renal and urinary disorders) | 0 | 0 | 0 | 1
Asthenia (General disorders) | 0 | 0 | 0 | 1
Near drowning (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Syncope (Nervous system disorders) | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Phase 1b Lead-in: Avelumab 800 mg + Pemetrexed/Carboplatin (N=6) | Phase 1b Lead-in: Avelumab 800 mg + Gemcitabine/Cisplatin (N=13) | Phase 1b Lead-in: Avelumab 1200 mg + Pemetrexed/Carboplatin (N=6) | Phase 1b and 2: Avelumab 1200 mg + Gemcitabine/Cisplatin (N=41)
Anaemia (Blood and lymphatic system disorders) | 3 | 10 | 1 | 26
Haemolytic anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
Leukopenia (Blood and lymphatic system disorders) | 0 | 2 | 0 | 6
Lymphopenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 3 | 8 | 4 | 23
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 4 | 4 | 20
Thrombocytosis (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 1 | 0 | 0
Intracardiac thrombus (Cardiac disorders) | 0 | 1 | 0 | 0
Palpitations (Cardiac disorders) | 0 | 1 | 0 | 0
Sinus bradycardia (Cardiac disorders) | 1 | 1 | 0 | 0
Tachycardia (Cardiac disorders) | 0 | 1 | 0 | 1
Tinnitus (Ear and labyrinth disorders) | 1 | 2 | 0 | 4
Hyperthyroidism (Endocrine disorders) | 0 | 1 | 0 | 1
Hypophysitis (Endocrine disorders) | 1 | 0 | 0 | 0
Hypothyroidism (Endocrine disorders) | 1 | 1 | 1 | 0
Conjunctival haemorrhage (Eye disorders) | 0 | 0 | 1 | 0
Dry eye (Eye disorders) | 1 | 0 | 0 | 0
Abdominal discomfort (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 2 | 4 | 0 | 3
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1 | 0 | 3
Abdominal rigidity (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Ascites (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 4 | 1 | 17
Diarrhoea (Gastrointestinal disorders) | 2 | 4 | 3 | 8
Dry mouth (Gastrointestinal disorders) | 1 | 2 | 0 | 2
Dyspepsia (Gastrointestinal disorders) | 0 | 4 | 0 | 3
Gastritis (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Gastrointestinal disorder (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 0 | 5
Glossodynia (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Lip dry (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Melaena (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 3 | 9 | 4 | 19
Oral disorder (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Pancreatic failure (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 1 | 0 | 0 | 2
Vomiting (Gastrointestinal disorders) | 1 | 5 | 1 | 14
Hepatitis (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Cytokine release syndrome (Immune system disorders) | 0 | 0 | 1 | 0
Candida infection (Infections and infestations) | 0 | 1 | 0 | 1
Cellulitis (Infections and infestations) | 1 | 0 | 0 | 0
Clostridium difficile infection (Infections and infestations) | 0 | 0 | 1 | 0
Conjunctivitis (Infections and infestations) | 1 | 0 | 0 | 1
Herpes zoster (Infections and infestations) | 0 | 1 | 0 | 0
Localised infection (Infections and infestations) | 0 | 1 | 0 | 0
Mucosal infection (Infections and infestations) | 1 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 0 | 1 | 0 | 1
Oral candidiasis (Infections and infestations) | 1 | 0 | 0 | 1
Oral herpes (Infections and infestations) | 1 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 1 | 0
Sepsis (Infections and infestations) | 1 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 2 | 1 | 0 | 1
Urinary tract infection (Infections and infestations) | 2 | 1 | 1 | 6
Urosepsis (Infections and infestations) | 0 | 1 | 0 | 0
Viral upper respiratory tract infection (Infections and infestations) | 0 | 0 | 1 | 0
Back injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 3
Fall (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 3
Femur fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1
Pelvic fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Procedural pneumothorax (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Skin abrasion (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Urinary tract stoma complication (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Alanine aminotransferase increased (Investigations) | 2 | 1 | 1 | 13
Amylase increased (Investigations) | 2 | 2 | 0 | 3
Aspartate aminotransferase increased (Investigations) | 2 | 1 | 0 | 9
Blood alkaline phosphatase increased (Investigations) | 0 | 1 | 0 | 8
Blood bilirubin increased (Investigations) | 0 | 1 | 0 | 2
Blood calcium increased (Investigations) | 0 | 1 | 0 | 0
Blood cholesterol increased (Investigations) | 0 | 1 | 0 | 3
Blood creatinine increased (Investigations) | 3 | 2 | 0 | 13
Blood pressure increased (Investigations) | 0 | 2 | 0 | 1
Blood thyroid stimulating hormone increased (Investigations) | 1 | 0 | 0 | 2
Blood triglycerides increased (Investigations) | 0 | 2 | 0 | 0
Body temperature increased (Investigations) | 0 | 1 | 0 | 0
Gamma-glutamyltransferase increased (Investigations) | 0 | 0 | 0 | 7
Haemoglobin decreased (Investigations) | 0 | 0 | 0 | 4
Lipase increased (Investigations) | 0 | 2 | 1 | 2
Lymphocyte count decreased (Investigations) | 0 | 3 | 0 | 1
Neutrophil count decreased (Investigations) | 0 | 3 | 0 | 5
Platelet count decreased (Investigations) | 4 | 4 | 1 | 9
Prothrombin time prolonged (Investigations) | 0 | 1 | 0 | 0
Troponin increased (Investigations) | 0 | 1 | 0 | 0
Weight decreased (Investigations) | 0 | 2 | 2 | 7
White blood cell count decreased (Investigations) | 2 | 3 | 0 | 6
Decreased appetite (Metabolism and nutrition disorders) | 2 | 3 | 1 | 11
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 2
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 1 | 0 | 3
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 2
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 1 | 1 | 0 | 4
Hyperuricaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 1
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 2 | 0 | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 2
Hypochloraemia (Metabolism and nutrition disorders) | 1 | 0 | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 2 | 1 | 0 | 5
Hypomagnesaemia (Metabolism and nutrition disorders) | 2 | 2 | 0 | 4
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1 | 1 | 4
Hypophosphataemia (Metabolism and nutrition disorders) | 3 | 0 | 0 | 2
Increased appetite (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 2 | 1 | 9
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 7
Chondropathy (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0 | 0
Clubbing (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Groin pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Myositis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Osteolysis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Spinal pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Ataxia (Nervous system disorders) | 0 | 1 | 0 | 1
Cognitive disorder (Nervous system disorders) | 1 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 6
Dizziness postural (Nervous system disorders) | 0 | 1 | 0 | 0
Dysgeusia (Nervous system disorders) | 1 | 2 | 0 | 5
Headache (Nervous system disorders) | 1 | 1 | 1 | 2
Hypoaesthesia (Nervous system disorders) | 0 | 1 | 0 | 2
Lethargy (Nervous system disorders) | 0 | 1 | 0 | 0
Neuralgia (Nervous system disorders) | 0 | 0 | 1 | 1
Neuropathy peripheral (Nervous system disorders) | 0 | 0 | 0 | 3
Presyncope (Nervous system disorders) | 0 | 1 | 0 | 1
Sciatica (Nervous system disorders) | 1 | 1 | 0 | 0
Taste disorder (Nervous system disorders) | 0 | 1 | 0 | 0
Tremor (Nervous system disorders) | 1 | 1 | 0 | 0
Agitation (Psychiatric disorders) | 0 | 1 | 0 | 2
Depression (Psychiatric disorders) | 0 | 0 | 0 | 3
Insomnia (Psychiatric disorders) | 2 | 1 | 0 | 1
Irritability (Psychiatric disorders) | 0 | 1 | 0 | 0
Mood altered (Psychiatric disorders) | 0 | 1 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 2 | 0 | 3
Chronic kidney disease (Renal and urinary disorders) | 0 | 1 | 0 | 1
Genitourinary symptom (Renal and urinary disorders) | 0 | 1 | 0 | 0
Haematuria (Renal and urinary disorders) | 0 | 3 | 0 | 2
Polyuria (Renal and urinary disorders) | 1 | 0 | 0 | 0
Renal impairment (Renal and urinary disorders) | 0 | 1 | 0 | 1
Urine odour abnormal (Renal and urinary disorders) | 0 | 1 | 0 | 0
Pelvic pain (Reproductive system and breast disorders) | 0 | 0 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 1 | 4
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 2 | 6
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 0 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 4
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 2 | 0 | 0
Dermal cyst (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 1 | 1 | 3
Erythema (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 1 | 0 | 4
Psoriasis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 3 | 1 | 5
Rash pruritic (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 0
Skin exfoliation (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 1 | 0 | 2
Hypertension (Vascular disorders) | 0 | 0 | 0 | 6
Lymphoedema (Vascular disorders) | 0 | 1 | 0 | 1
Superficial vein thrombosis (Vascular disorders) | 0 | 1 | 0 | 1
Thrombosis (Vascular disorders) | 0 | 1 | 0 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 3
Asthenia (General disorders) | 2 | 2 | 0 | 11
Chest pain (General disorders) | 1 | 0 | 1 | 1
Discomfort (General disorders) | 0 | 1 | 0 | 0
Extravasation (General disorders) | 0 | 1 | 0 | 0
Fatigue (General disorders) | 3 | 8 | 3 | 15
Influenza like illness (General disorders) | 1 | 2 | 0 | 1
Mucosal inflammation (General disorders) | 1 | 0 | 0 | 1
Oedema peripheral (General disorders) | 0 | 2 | 0 | 3
Pain (General disorders) | 0 | 1 | 0 | 3
Pyrexia (General disorders) | 2 | 1 | 0 | 11
Thirst (General disorders) | 0 | 1 | 0 | 0
Chills (General disorders) | 0 | 0 | 0 | 3
Hypertransaminasaemia (Hepatobiliary disorders) | 1 | 1 | 0 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Influenza (Infections and infestations) | 0 | 1 | 0 | 0
Rhinitis (Infections and infestations) | 0 | 1 | 0 | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 0 | 3

LIMITATIONS AND CAVEATS:
The study was terminated since there was no need for further safety or efficacy data to be collected. The subjects having benefit from the investigational treatments have been moved to a continuation study NCT05059522

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2018-10-02): https://cdn.clinicaltrials.gov/large-docs/96/NCT03317496/Prot_000.pdf
  • Statistical Analysis Plan (2021-02-10): https://cdn.clinicaltrials.gov/large-docs/96/NCT03317496/SAP_001.pdf